CLINICAL TRIAL: NCT07279974
Title: The Effect of Preoperative Video-Based Education on Fear of Mobilization in Patients Undergoing Total Hip Arthroplasty: A Randomized Controlled Trial
Brief Title: Preoperative Video-Based Education in Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Nermin Ocaktan, assistant professor, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-17-46
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Total Hip Arthroplasty (THA); Kinesiophobia; Postoperative Pain; Early Mobilization; Hip Osteoarthritis; Musculoskeletal Rehabilitation
Keywords: Total Hip Arthroplasty; Kinesiophobia; Fear of Movement; Preoperative Education; Video-Based Training; Mobilization; Postoperative Pain; Rehabilitation Nursing; Orthopedic Surgery; Early Mobilization
MeSH Terms: conditions — Kinesiophobia; Pain, Postoperative; Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment design in which participants are randomly allocated to either an intervention group receiving preoperative video-based mobilization education or a control group receiving standard verbal education. Both groups are followed concurrently, and no crossover occurs between groups. Outcomes are assessed on the first postoperative day.
Masking Description: Due to the nature of the intervention (video-based education), neither participants nor care providers could be blinded. Outcome assessment was conducted by a researcher who was not involved in randomization; however, full blinding was not feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this arm receive routine preoperative verbal education plus a structured video-based mobilization training. The video includes demonstrations of bed exercises, mobilization with assistive devices, chair transfer techniques, toilet use, stair negotiation, and postoperative precautions.
  Interventions: Behavioral: Video-Based Mobilization Education
- Control Group (Active Comparator): Participants in this arm receive only routine preoperative verbal education provided by ward nurses. No video-based training is given.
  Interventions: Behavioral: Standard Verbal Education

INTERVENTIONS:
Behavioral: Video-Based Mobilization Education — A structured preoperative video-based mobilization training including demonstrations of bed exercises, mobilization with assistive devices, chair transfer, toilet use, stair negotiation, and postoperative precautions.
  Arms: Intervention Group
Behavioral: Standard Verbal Education — Routine preoperative verbal instruction provided by ward nurses.
  Arms: Control Group

SUMMARY:
This single-center, prospective, randomized controlled trial aims to evaluate the effect of preoperative video-based mobilization education on postoperative fear of movement (kinesiophobia), pain during first mobilization, and early mobilization characteristics in patients undergoing total hip arthroplasty. Ninety-six participants were randomized to receive either routine verbal education plus video-based education or routine verbal education alone. Postoperative outcomes were assessed using the Tampa Scale of Kinesiophobia (TSK), Numerical Pain Rating Scale (NPRS), and standardized mobilization observation forms.

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) is a common orthopedic procedure in which early postoperative mobilization plays a key role in preventing complications, reducing pain, and accelerating functional recovery. However, fear of movement (kinesiophobia), insufficient preoperative preparation, and uncertainty regarding mobility expectations may negatively affect patients' early rehabilitation performance. Providing structured, standardized education before surgery has been shown to improve postoperative participation and enhance patient confidence, yet the most effective format of such education remains unclear.

This randomized controlled trial was designed to evaluate the impact of a preoperative video-based mobilization education program on postoperative kinesiophobia, pain during the first mobilization, and early mobilization characteristics among patients undergoing primary THA. A total of 96 participants were randomly assigned to an intervention group or a control group using a simple randomization method. Both groups received routine preoperative verbal education, while the intervention group additionally viewed a structured mobilization training video developed by a multidisciplinary team of orthopedic surgeons, physiatrists, physiotherapists, and orthopedic nurses.

The educational video included demonstrations of bed exercises, safe ambulation techniques with assistive devices, chair transfer mechanics, toilet use, stair negotiation, and postoperative precautions. All postoperative outcomes were measured on the first postoperative day following each patient's initial mobilization session. Kinesiophobia was assessed using the Tampa Scale of Kinesiophobia (TSK); pain intensity was measured using the Numerical Pain Rating Scale (NPRS) immediately before and after the first mobilization; and mobilization characteristics (duration, number of steps, activity level, and level of assistance required) were recorded using a standardized observation form.

The aim of the study was to determine whether video-based preoperative education provides measurable benefits compared with routine verbal instruction alone. By focusing on both psychological (kinesiophobia) and physical (pain and mobilization performance) outcomes, this trial seeks to contribute new evidence to the field of musculoskeletal rehabilitation and to support more effective perioperative education strategies in THA care. No adverse events related to the intervention were reported.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years or older

Able to communicate verbally

Scheduled for primary total hip arthroplasty

No major neurological disease

No major psychiatric disease

Able to participate in postoperative mobilization

Provided written informed consent

Exclusion Criteria:

Scheduled for revision total hip arthroplasty

Comorbidities that prevent safe mobilization (e.g., severe cardiopulmonary limitations, severe balance disorders)

Severe cognitive impairment affecting comprehension or cooperation

Any condition preventing participation in the mobilization protocol

Declining to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Kinesiophobia (TSK Score) | First postoperative day, after first mobilization
  Kinesiophobia will be measured using the Tampa Scale of Kinesiophobia (TSK), a 17-item scale scored on a 4-point Likert system (1-4). Total scores range from 17 to 68, with higher scores indicating greater fear of movement. The Turkish validated version will be used.

SECONDARY OUTCOMES:
Pain Intensity Before First Mobilization | Immediately before first mobilization
  Pain intensity will be assessed using the Numerical Pain Rating Scale (NPRS), in which patients rate their pain on a scale from 1 to 10. Higher scores represent greater pain intensity.
Pain Intensity After First Mobilization | Immediately after first mobilization
  Pain intensity will be assessed using the Numerical Pain Rating Scale (NPRS), recorded on a scale from 1 to 10, where higher scores indicate more severe pain.
Mobilization Duration | First postoperative day
  The total duration (in minutes) of the patient's first mobilization session will be recorded by the researcher using a standardized observation form.
Number of Steps During First Mobilization | First postoperative day
  The number of steps taken during the first mobilization session will be counted using the standardized mobilization observation form.
Activity Level During First Mobilization | First postoperative day
  Activity level will be evaluated using the standardized mobilization observation form, which records walking distance, device use, and functional quality of ambulation.
Level of Assistance Required During First Mobilization | First postoperative day
  The required level of assistance (independent, minimal assistance, moderate assistance, or full assistance) will be assessed during the first mobilization session using a standardized observation form.

CONTACTS AND LOCATIONS:
Overall Officials: Nermin Ocaktan, Principal Investigator — Acıbadem Mehmet Ali Aydınlar University
Locations (1):
- Acibadem Healthcare Group Hospital - Orthopedic Clinic, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared because the study does not include a data sharing provision in the ethics approval and the collected data contain potentially identifiable clinical information.